CLINICAL TRIAL: NCT01812265
Title: A Double Blind (3rd Party Open), Randomized, Placebo Controlled, Crossover Study To Investigate The Effects Of Pf-06305591 On Cold Pain In Healthy Male Subjects
Brief Title: Cold Pressor Test is Used in This Study to Assess the Effect of PF-06305591 on Pain Intensity Evoked by Cold in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B5281003
Record Dates: First submitted 2013-03-11; First posted 2013-03-18 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- PF-06305591 Dose 1 (Experimental)
  Interventions: Drug: PF-06305591
- PF-06305591 Dose 2 (Experimental)
  Interventions: Drug: PF-06305591
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06305591 — single Dose
  Arms: PF-06305591 Dose 1
Drug: PF-06305591 — single Dose
  Arms: PF-06305591 Dose 2
Drug: Placebo — Single Dose
  Arms: Placebo

SUMMARY:
This study will evaluate the pharmacological activity of PF-06305591 in healthy male volunteers by assessing the effects of two dose levels of PF-06305591 on cold pain intensity evoked by keeping non-dominant hand into a water bath kept at 2+/- degrees.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Subjects unable to tolerate pre-study Cpressor testing at screening.
* Subjects with an average pain (AUC 0 to 120 sec) in the pre-study Cpressor test of less than or equal to 20.
* Broken skin on hands or forearms

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Visual Analogue Scale (VAS) Score at time X, measured within a 2 minute interval | 24h
  Change from Baseline in 10 cm VAS pain score; 10-point pain intensity ordinal rating system: 0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = worst possible pain. Change = scores at observation minus score at Baseline in a 2 minute assessment.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 24h
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5281003&StudyName=Cold%20Pressor%20test%20is%20used%20in%20this%20study%20to%20assess%20the%20effect%20of%20PF-06305591%20on%20pain%20intensity%20evoked%20by%20cold%20in%20Healthy%20Male%20Sub